CLINICAL TRIAL: NCT00027508
Title: Phase II Study Of ET-743 In Patients With Unresectable Malignant Pleural Mesothelioma
Brief Title: Ecteinascidin 743 in Treating Patients With Malignant Mesothelioma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Enrolment halted prematurely and not resumed. 2 patients enrolled. No data was obtained.
Sponsor: PharmaMar (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: MSKCC-01084; CDR0000069034 (Registry Identifier: PDQ (Physician Data Query)); PMAR-ET-B-020-99; NCI-G01-2026
Record Dates: First submitted 2001-12-07; First posted 2004-01-15 (Estimated); Last update posted 2015-02-24 (Estimated); Status verified 2013-06

CONDITIONS: Malignant Mesothelioma
Keywords: advanced malignant mesothelioma; recurrent malignant mesothelioma
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Trabectedin

INTERVENTIONS:
Drug: trabectedin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of ecteinascidin 743 in treating patients who have malignant mesothelioma that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine partial and complete response rates in patients with unresectable malignant mesothelioma treated with ecteinascidin 743. II. Determine the toxicity profile of this drug in these patients. III. Determine the pharmacokinetic/pharmacodynamic relationships of this drug in these patients. IV. Determine the duration of response, time to disease progression, 6-month progression-free survival, time to treatment failure, and overall survival of patients treated with this drug. V. Assess the quality of life of these patients treated with this drug.

OUTLINE: This is a multicenter study. Patients receive ecteinascidin 743 IV over 3 hours on day 1. Treatment repeats every 3 weeks for at least 6 courses in the absence of disease progression or unacceptable toxicity. Patients with a complete response (CR) receive 2 additional courses after achieving CR. Quality of life is assessed at baseline and at the beginning of each course of therapy. Patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 20-36 patients will be accrued for this study within 12-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed malignant mesothelioma that is not amenable to curative surgery At least 1 unidimensionally measurable lesion that is at least 15 mm by CT scan OR At least 1 bidimensionally measurable lesion that is at least 10 mm by CT scan Lesions in previously irradiated area are not considered measurable unless there is evidence of progression No symptomatic brain or leptomeningeal involvement

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-1 OR Karnofsky 70-100% Life expectancy: At least 3 months Hematopoietic: Neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 10 g/dL Hepatic: Bilirubin no greater than upper limit of normal (ULN) Alkaline phosphatase no greater than ULN unless bone metastases are present AST/ALT no greater than 2.5 times ULN Albumin at least 2.5 g/dL No chronic active liver disease Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 40 mL/min Cardiovascular: No uncontrolled heart disease No uncontrolled hypertension Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception during and for one month after study No other serious illness or medical condition No history of significant neurological or psychiatric disorders No significant active infection No other concurrent neoplastic disease except non-melanoma skin cancer or carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: No prophylactic hematopoietic colony-stimulating factors (e.g., filgrastim (G-CSF) or sargramostim (GM-CSF)) Chemotherapy: No prior systemic chemotherapy No other concurrent chemotherapy Endocrine therapy: No concurrent hormonal therapy Radiotherapy: See Disease Characteristics At least 30 days since prior radiotherapy and recovered No concurrent radiotherapy except palliative local radiotherapy to non-target lesions Surgery: See Disease Characteristics At least 14 days since prior pleurodesis Recovered from prior surgery Other: At least 30 days since prior participation in another therapeutic clinical trial or therapy with other investigational drugs No concurrent treatment for other neoplastic disease No other concurrent experimental anticancer medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-07; Primary Completion 2002-02 (Actual); Study Completion 2002-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee M. Krug, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (4):
- United States (4):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan-Kettering Cancer Center, New York, New York